CLINICAL TRIAL: NCT03343613
Title: A Phase 1a/1b Study of an Anti-IDO-1 Agent (LY3381916) Administered Alone or in Combination With Anti- PD-L1 Checkpoint Antibody (LY3300054) in Solid Tumors
Brief Title: A Study of LY3381916 Alone or in Combination With LY3300054 in Participants With Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due to strategic business decision by Eli Lilly and Company.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16786; I9L-MC-JZCA (Other: Eli Lilly and Company); 2017-002693-39 (EudraCT Number)
Record Dates: First submitted 2017-11-09; First posted 2017-11-17 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Solid Tumor; Non Small Cell Lung Cancer; Renal Cell Carcinoma; Triple Negative Breast Cancer
Keywords: IDO-1 Inhibitor; IDO1 Inhibitor; IDO Inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Triple Negative Breast Neoplasms | interventions — IDO-1 inhibitor LY3381916; LY3300054

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- LY3381916 Escalation (Experimental): LY3381916 administered orally.
  Interventions: Drug: LY3381916
- LY3381916 + LY3300054 Escalation (Experimental): LY3381916 administered orally and LY3300054 administered intravenously (IV).
  Interventions: Drug: LY3381916; Drug: LY3300054
- LY3381916 Expansion (Experimental): LY3381916 administered orally.
  Interventions: Drug: LY3381916
- LY3381916 + LY3300054 Expansion B1 (Experimental): Metastatic triple negative breast cancer (TNBC)
  LY3381916 administered orally and LY3300054 administered IV.
  Interventions: Drug: LY3381916; Drug: LY3300054
- LY3381916 + LY3300054 Expansion B2 (Experimental): Metastatic non-small cell lung cancer (NSCLC)
  LY3381916 administered orally and LY3300054 administered IV.
  Interventions: Drug: LY3381916; Drug: LY3300054
- LY3381916 + LY3300054 Expansion B3 (Experimental): Metastatic clear cell carcinoma renal cell carcinoma (RCC)
  LY3381916 administered orally and LY3300054 administered IV.
  Interventions: Drug: LY3381916; Drug: LY3300054

INTERVENTIONS:
Drug: LY3381916 — IDO-1 inhibitor administered orally
Drug: LY3300054 — PD-L1 inhibitor administered IV
  Arms: LY3381916 + LY3300054 Escalation; LY3381916 + LY3300054 Expansion B1; LY3381916 + LY3300054 Expansion B2; LY3381916 + LY3300054 Expansion B3

SUMMARY:
The purpose of this study is to evaluate the safety of the study drug LY3381916 administered alone or in combination with anti-programmed cell death ligand 1 (PD-L1) checkpoint antibody (LY3300054).

ELIGIBILITY:
Inclusion Criteria:

* Dose escalation phase: Participant must have histological or cytological evidence of a diagnosis of cancer that is advanced and/or metastatic.
* Dose expansion B1: Metastatic TNBC participants who have not received prior PD-1/L1 treatment.
* Dose expansion B2: Metastatic NSCLC participants who have progressed on prior PD-L1/L1 treatment.
* Dose expansion B3: Metastatic clear cell carcinoma RCC who have progressed on prior PD-L1/L1 treatment.
* Have adequate organ function.
* Have a performance status (PS) of ≤1 on the Eastern Cooperative Oncology Group (ECOG) scale.
* Are able and willing to provide required, newly acquired tumor biopsies.
* Have discontinued previous treatments for cancer.
* Are able to swallow capsules.

Exclusion Criteria:

* Currently enrolled in a clinical study.
* Have known symptomatic central nervous system metastases or carcinomatous meningitis.
* Have a serious concomitant systemic disorder.
* Have a symptomatic human immunodeficiency virus infection or symptomatic activated/reactivated hepatitis B or C.
* Have a significant cardiac condition.
* Have previously received an indoleamine- 2,3-dioxygenase (IDO) inhibitor.
* Have an active autoimmune disease or currently require immunosuppression of >10 milligrams of prednisone or equivalent per day.
* Have interstitial lung disease or (noninfectious) pneumonitis, participants with a history of (noninfectious) pneumonitis that required steroids to assist with management.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-05-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities (DLTs) | Baseline through Cycle 1 (28 Day Cycle)
  Number of participants with DLTs

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Plasma Concentration (Cmax) of LY3381916 | Predose Lead in Day 1 through Cycle 3 Day 1
  PK: Cmax of LY3381916
PK: Area Under the Plasma Concentration Curve (AUC) of LY3381916 | Predose Lead in Day 1 through Cycle 3 Day 1
  PK: AUC of LY3381916
PK: Cmax of LY3381916 Administered in Combination with LY3300054 | Predose Cycle 1 Day 1 through Cycle 3 Day 1
  PK: Cmax of LY3381916 administered in combination with LY3300054
PK: AUC of LY3381916 Administered in Combination with LY3300054 | Predose Cycle 1 Day 1 through Cycle 3 Day 1
  PK: AUC of LY3381916 administered in combination with LY3300054
PK: Cmax of LY3300054 Administered in Combination with LY3381916 | Predose Cycle 1 Day 1 through Cycle 3 Day 1
  PK: Cmax of LY3300054 administered in combination with LY3381916
PK: Minimum Plasma Concentration (Cmin) of LY3300054 Administered in Combination with LY3381916 | Predose Cycle 1 Day 1 through Cycle 3 Day 1
  PK: Cmin of LY3300054 administered in combination with LY3381916
Objective Response Rate (ORR): Percentage of Participants with a Complete Response (CR) or Partial Response (PR) | Baseline through Measured Progressive Disease (Estimated up to 12 Months)
  ORR: Percentage of participants with a CR or PR
Time to Response (TTR) | Baseline to Date of CR or PR (Estimated up to 12 Months)
  TTR
Disease Control Rate (DCR): Percentage of Participants who Exhibit Stable Disease (SD), CR or PR | Baseline through Measured Progressive Disease (Estimated up to 12 Months)
  DCR: Percentage of participants who exhibit SD, CR or PR
Duration of Response (DOR) | Date of CR or PR to Date of Objective Progression or Death Due to Any Cause (Estimated up to 12 Months)
  DOR
Progression Free Survival (PFS) | Baseline to Objective Progression or Death Due to Any Cause (Estimated Up to 12 Months)
  PFS

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (12):
- United States (3):
  - IU Simon Cancer Center, Indianapolis, Indiana
  - Sarah Cannon Research Institute SCRI, Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
- Belgium (3):
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
- Finsen Institute, Copenhagen, Denmark
- Gustave Roussy, Villejuif, France
- Italy (2):
  - Azienda Ospedaliera San Gerardo, Monza, Milano
  - Azienda Ospedaliera Umberto I, Ancona
- Spain (2):
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga, Andalusia
  - Hospital Universitari Vall d'Hebron, Barcelona

REFERENCES:
- See also: A Study of LY3381916 Alone or in Combination With LY3300054 in Participants With Solid Tumors — https://trials.lillytrialguide.com/en-US/trial/5sqQ8KzLnN79i471hIpC0c?conditionId=LcQNUbMtMWSEYwOSaGUIi